CLINICAL TRIAL: NCT04611880
Title: A Trial of Crizanlizumab for the Treatment of Retinal Vasculopathy With Cerebral Leukoencephalopathy (RVCL)
Brief Title: Crizanlizumab for Treatment of Retinal Vasculopathy With Cerebral Leukoencephalopathy (RVCL)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202008079
Record Dates: First submitted 2020-10-26; First posted 2020-11-02 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: RVCL - Retinal Vasculopathy Cerebral Leukoencephalopathy
MeSH Terms: conditions — Vasculopathy, Retinal, With Cerebral Leukodystrophy | interventions — crizanlizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm Study (Other): Single arm study: crizanlizumab will be supplied in single use vials containing 10 mL at a concentration of 10 mg/mL for administration by IV infusion. Each patient will receive one dose of crizanlizumab on day 1 of Week 1, day 1 of Week 3, day 1 of Week 7, and then day 1 of every 4-week cycle. On infusion day, the pharmacist or designated personnel will prepare individual doses of crizanlizumab for subjects on a milligram per kilogram basis (5 mg/kg) in a 100 mL infusion bag in accordance with the Pharmacy Manual. Crizanlizumab will be administered over 30 minutes by IV infusion
  Interventions: Drug: Crizanlizumab

INTERVENTIONS:
Drug: Crizanlizumab — Drug: crizanlizumab is a humanized monoclonal anti-P-selectin antibody that prevents leukocyte adhesion to the vascular endothelium, thereby limiting risk of microvascular occlusion. It is administered intravenously.
  Other Names: ADAKVEO

SUMMARY:
This is a Phase 2 trial that will test the efficacy and safety of crizanlizumab for the treatment of retinal vasculopathy with cerebral leukoencephalopathy (RVCL), a very rare and uniformly fatal genetic condition that affects the microvasculature, especially of the brain and eye. There currently is no treatment for RVCL. A maximum of 20 patients will be enrolled.

DETAILED DESCRIPTION:
Retinal vasculopathy with cerebral leukoencephalopathy (RVCL) is a very rare and uniformly fatal genetic condition that affects the microvasculature, especially of the brain and eye. Symptoms begin in adulthood (usually in the mid-30s to early 40s) and include loss of vision, mini-strokes, and dementia. Other patients have suffered from microvascular disease involving the kidneys, osteonecrosis, and gut ischemia. Some of these features of microvascular occlusive disease resemble ischemic events that occur during sickle cell disease. Currently, there is no effective treatment for RVCL.

The goal of this study is to test the efficacy of RVCL patients treated with crizanlizumab, a humanized monoclonal anti-P-selectin antibody that prevents leukocyte adhesion to the vascular endothelium, thereby limiting risk of microvascular occlusion. P-selectin is mobilized to the surface of activated vascular endothelial cells and promotes leukocyte adhesion to the blood vessel wall. The Miner laboratory has preliminarily observed a correlation with levels of soluble P-selectin and the number of brain lesions in patients with RVCL. Since leukocyte adhesion to the vascular endothelium promotes microvascular occlusion, we will determine if crizanlizumab will help to limit ischemia and brain lesions in patients with RVCL. This may lead to the development of fewer ischemic brain and eye lesions.

Up to 20 RVCL patients will receive intravenous infusions of crizanlizumab 5 mg/kg at weeks 1 and 3. Thereafter, patients will receive crizanlizumab 5 mg/kg every 28 days for a total of 24 total months. Monitoring will include standard-of-care serial MRI as well as standard-of-care eye disease monitoring at pre-defined intervals. High-risk medication monitoring will include blood work monitoring (CBC/CMP) 1 month after initiation of treatment and every 3 months thereafter. Standard-of-care assessments will be performed including radiological and physical examinations as well as eye imaging and examinations. Patients will be followed for at least 2 years after completion of crizanlizumab administration.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of RVCL with confirmation by genetic test
2. At least 25 years of age with imaging evidence of brain or eye disease at the time of study registration
3. Normal hematologic function defined as: White blood cell count (WBC) > 4x109/L, Absolute neutrophil count (ANC) >1.5x109/L and Platelets > 100x109/L
4. Females of childbearing potential (FCBP) must agree to refrain from becoming pregnant while on study drug and for 3 months after discontinuation from study drug, and must agree to use adequate contraception including hormonal contraception, (i.e. birth control pills, etc), barrier method contraception (i.e. condoms), or abstinence during that time-frame
5. Able to understand and willing to sign an Internal Review Board (IRB)-approved written informed consent document (or that of legally authorized representative, if applicable)

   -

Exclusion Criteria:

1. Acute bacterial, fungal, or viral infection
2. Known HIV, untreated latent tuberculosis (TB), or active hepatitis B or C infection or zoster
3. Pregnant and/or breastfeeding. Negative serum pregnancy test required prior to starting study treatment. For females of child-bearing potential (FCBP), a negative urine pregnancy test is required before each infusion.
4. Known hypersensitivity to one or more of the study agents
5. Currently receiving or has received any investigational drugs within the 14 days prior to the first dose of study drug
6. Liver function tests (LFTs) higher than 3x the upper limit of normal within the last 30 days
7. Treatment with other monoclonal antibody medications within the last 30 days
8. Treatment with various forms of anticoagulation within last 30 days, including but not limited to clopidogrel or coumadin or direct thrombin inhibitors

   -

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-01-25 (Actual); Primary Completion 2025-04-02 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in lesion pattern on Fluid-Attenuated Inversion Recovery (FLAIR) Magnetic Resonance Imaging (MRI) in RVCL patients. | year
  Volume change in lesions of FLAIR MRI between baseline and one year is assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Andria Ford, MD, Principal Investigator — Washington University School of Medicine
Locations (2):
- United States (2):
  - Andria Ford, St Louis, Missouri
  - Perelman School of Medicine; University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared among the principle investigator and the other investigators
Supporting Information: Study Protocol, ICF
Time Frame: immediate
Access Criteria: Individual Patient Data (IPD) will be available on REDCap or as provided by principal investigator

REFERENCES:
- [Background] Kavanagh D, Spitzer D, Kothari PH, Shaikh A, Liszewski MK, Richards A, Atkinson JP. New roles for the major human 3'-5' exonuclease TREX1 in human disease. Cell Cycle. 2008 Jun 15;7(12):1718-25. doi: 10.4161/cc.7.12.6162. Epub 2008 Jun 16. PMID 18583934
- [Background] Hasan M, Fermaintt CS, Gao N, Sakai T, Miyazaki T, Jiang S, Li QZ, Atkinson JP, Morse HC 3rd, Lehrman MA, Yan N. Cytosolic Nuclease TREX1 Regulates Oligosaccharyltransferase Activity Independent of Nuclease Activity to Suppress Immune Activation. Immunity. 2015 Sep 15;43(3):463-74. doi: 10.1016/j.immuni.2015.07.022. Epub 2015 Aug 25. PMID 26320659
- [Background] Wood KC, Hebbel RP, Granger DN. Endothelial cell P-selectin mediates a proinflammatory and prothrombogenic phenotype in cerebral venules of sickle cell transgenic mice. Am J Physiol Heart Circ Physiol. 2004 May;286(5):H1608-14. doi: 10.1152/ajpheart.01056.2003. Epub 2004 Jan 2. PMID 14704223
- [Background] McEver RP, Cummings RD. Role of PSGL-1 binding to selectins in leukocyte recruitment. J Clin Invest. 1997 Dec 1;100(11 Suppl):S97-103. No abstract available. PMID 9413410
- [Background] Ford AL, Chin VW, Fellah S, Binkley MM, Bodin AM, Balasetti V, Taiwo Y, Kang P, Lin D, Jen JC, Grand MG, Bogacki M, Liszewski MK, Hourcade D, Chen Y, Hassenstab J, Lee JM, An H, Miner JJ, Atkinson JP. Lesion evolution and neurodegeneration in RVCL-S: A monogenic microvasculopathy. Neurology. 2020 Oct 6;95(14):e1918-e1931. doi: 10.1212/WNL.0000000000010659. Epub 2020 Sep 4. PMID 32887784
- [Derived] Wang WX, Spiegelman D, Rao PK, Rhee RL, Ford AL, Miner JJ, Apte RS. Crizanlizumab for retinal vasculopathy with cerebral leukoencephalopathy in a phase II clinical study. J Clin Invest. 2024 May 7;134(12):e180916. doi: 10.1172/JCI180916. PMID 38950286
- See also: RVCL Research and Treatment Center — http://rvcl-research.wustl.edu